CLINICAL TRIAL: NCT06181682
Title: Intranasal Dexmedetomidine Versus Intranasal Midazolam as a Premedication in Pediatrics Undergoing Upper GI Endoscopy
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Marwa Mostafa Hasan Salem, Principal Investigator, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: ASU MS
Record Dates: First submitted 2023-12-10; First posted 2023-12-26 (Actual); Last update posted 2023-12-26 (Actual); Status verified 2023-12

CONDITIONS: Anesthesia
MeSH Terms: interventions — Dexmedetomidine; Midazolam

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- dexmedetomidine group (Active Comparator): patients will receive intranasal dexmedetomidine (1 microgram/kg) -Intranasal dexmedetomidine will be prepared from the 100 mcg/ml parenteral preparation in a 1-ml syringe, and 0.9% saline will be added to make a final volume of 1 ml- (0.5 ml will be administrated in each nostril) before starting the anesthesia with monitoring of sedation level and oxygen saturation.
  Interventions: Drug: Dexmedetomidine
- midazolam group (Active Comparator): patients will receive intranasal midazolam (0.2 mg/kg) up to 5 mg - Intranasal midazolam will be prepared from a 5 mg/ml parenteral preparation, and 0.9% saline will be added to make a final volume of one ml in a 1-ml syringe- (0.5 ml will be administrated in each nostril) before starting the anesthesia with monitoring of sedation level and oxygen saturation.
  Interventions: Drug: Midazolam

INTERVENTIONS:
Drug: Dexmedetomidine — Intranasal Dexmedetomidine
  Other Names: Precedex
  Arms: dexmedetomidine group
Drug: Midazolam — Intranasal midazolam
  Other Names: Dormicum
  Arms: midazolam group

SUMMARY:
compare the effectiveness of intranasal dexmedetomidine and midazolam as a premedication in sedation of preschool children in GI endoscopy

ELIGIBILITY:
Inclusion Criteria:

* Children of preschool age (2-6 years old).
* American scocity of anaesthesiology (ASA) I - II children.
* Expected duration of the procedure is less than 50 minutes.

Exclusion Criteria:

* Cardiac arrhythmia, congenital heart disease, or hemodynamic or respiratory instability; children at risk for airway obstruction.
* Behavioral, mental or developmental abnormality (example: mental retardation, Attention Deficit Hyperactivity Disorder "ADHD", Autism, Down syndrome).
* Regular intake of either brain stimulant or depressive drugs (example: Methylphenidate, amphetamine-dextroamphetamine and diazepam respectively).
* Parent's refusal.
* Emergency case.
* Allergy to any of the used drugs

Ages: 2 Years to 6 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 70 (Estimated)
Dates: Start 2024-01 (Estimated); Primary Completion 2024-03 (Estimated); Study Completion 2024-03 (Estimated)

PRIMARY OUTCOMES:
Sedation status at separation from the parent | within 30 minutes after drugs administration
  Parental separation anxiety scale (PSAS) ,A score of 1-2 was considered "satisfactory separation" and a score of 3-4 was considered "unsatisfactory separation."

SECONDARY OUTCOMES:
Onset of sedation | within 30 minutes after drugs administration
  Onset of sedation will be recorded according to Modified RAMSAY Sedation Scale when the score reaches 3 points, patient is then ready to be transferred.
awakening time | within 15 minutes after end of anaesthesia
  recovery time (defined as return of consciousness, recovery of protective air way reflexes and resumption of motor activity)
post-operative emergence delirium and agitation. | within 30 minutes from recovery
  (PAED) scale: Pediatric Anesthesia Emergence Delirium (PAED) scales. scale from 0 to 20. higher scores mean a worse outcome